CLINICAL TRIAL: NCT06535152
Title: CLINIMARK Clinical Investigation Plan Lifelight Non-Invasive Blood Pressure Validation Study PR 2021-443
Brief Title: Lifelight Non-Invasive Blood Pressure and Heart Rate Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xim Limited (Industry)
Collaborators: Element Materials Technology (Industry); Mind Over Matter Medtech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PR 2021-443
Record Dates: First submitted 2024-07-18; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Up to eight pairs of reference and Lifelight recordings (starting and ending with reference recordings) were taken sequentially to obtain a minimum of three valid paired reference and Lifelight BP measurements. At least 60 seconds elapsed between each BP determination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifelight and BP measurement (Experimental): The accuracy of Lifelight's blood pressure measurements was assessed by comparing Lifelight's measurements with measurements made by dual-observer manual auscultation using the same-arm sequential method specified in ISO 81060-2:2018/AMD 1:2020. The accuracy of Lifelight's pulse rate measurements was assessed by comparing Lifelight's measurements with concurrent ECG-derived heart rate values. The participants were resting before their measurements were taken to ensure stable blood pressure. For each Lifelight measurement, two sets of blood pressure measurements were taken using dual-observer manual auscultation. The first measurement was taken before the Lifelight measurement and the second just after. If there was too much variation between the before and after measurement, or between the 2 independent observers, the measurement was discarded and repeated. For this validation procedure, the measurements taken during the original study were re-processed in the new updated algorithm.
  Interventions: Device: Lifelight; Device: Manual sphygmomanometer

INTERVENTIONS:
Device: Lifelight — Lifelight is a artificial-intelligence software application that enables completely contactless spot measurements (i.e., one-off measurements without prior calibration) of PR and BP. Based on the science of remote photoplethysmography (rPPG), Lifelight works by detecting tiny changes in the colour of facial skin that occur every time the heart beats. All that is required to generate PR and BP measurements is that the software application is downloaded onto a computer device (e.g., smartphone or tablet) with a standard camera, and that the patient's face stays in the line of sight of the camera for up to 60 seconds.
Device: Manual sphygmomanometer — Blood Pressure Measurement

SUMMARY:
Lifelight is a novel, calibration-free, software-only medical device that contactlessly measures pulse rate and blood pressure by measuring remote photoplethysmography (rPPG) signals of a patient's face using a standard smartphone or tablet camera.

By conducting this validation study we aimed to demonstrate the accuracy of Lifelight for classifying the full range of clinically relevant blood pressures as hypertensive or non-hypertensive and demonstrate its accuracy for measuring pulse rate and the blood pressure of people with blood pressures relevant to Stage 1 hypertension.

DETAILED DESCRIPTION:
Lifelight was investigated in a study that followed the data collection and data analysis methodology outlined in ISO 81060-2:2018/AMD 1:2020 "Non-invasive Sphygmomanometers - Part 2: Clinical investigation of automated measurement type". This validation study was conducted by independent laboratory Element Materials Technology Boulder (formerly Clinimark), a global leader for clinical testing of vital sign data for medical devices and consumer wearable products. The study generated data from 85 people aged 18-85 with the wide-ranging distribution of blood pressures specified in ISO 81060-2:2018/AMD 1:2020.The accuracy of Lifelight's blood pressure measurements was assessed by comparing Lifelight's measurements with measurements made by dual-observer manual auscultation using the same-arm sequential method specified in ISO 81060-2:2018/AMD 1:2020. The accuracy of Lifelight's pulse rate measurements was assessed by comparing Lifelight's measurements with concurrent ECG-derived heart rate values. Data was collected in an Independent Review Board-approved study conducted by independent laboratory Clinimark (now Element) in the USA and repurposed for the testing of the new improved model in the latest version of the Lifelight® EA device. The data collected consists of 85 participants, with three readings each. The participants were resting before their measurements were taken to ensure stable blood pressure. For each Lifelight measurement, two sets of blood pressure measurements were taken using dual-observer manual auscultation. The first measurement was taken before the Lifelight measurement and the second just after. If there was too much variation between the before and after measurement, or between the two independent observers, the measurement was discarded and repeated. For this validation procedure, the measurements taken during the original study were re-processed in the new updated algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 18 to 85 years old

Exclusion Criteria:

* Participants were excluded from the study if they were medically unsuitable for participation at time of visit, any heart dysrhythmias (except respiratory sinus arrhythmia) as confirmed with a 3 lead ECG, compromised circulation or peripheral vascular disease, clotting disorders, female participants who were pregnant or trying to get pregnant, excessive facial hair, and conditions that affect the skin, such as anaemia, jaundice, rosacea, psoriasis, acute acne, and erythropoietic protoporphyria.

Participants could choose to withdraw themselves from the study without prejudice or they could be withdrawn by study investigators for predetermined reasons. Data excluded from the analysis was documented with justifications.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-05-18 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Classification Accuracy | Up to 3 Months
  Demonstrate the accuracy of Lifelight for classifying the full range of clinically relevant blood pressures as hypertensive or non-hypertensive.
Pulse Rate Measurement Accuracy (relevant to Stage 1 hypertension | Up to 3 Months
  Demonstrate its accuracy for measuring pulse rate (bpm)
Blood Pressure Measurement Accuracy (relevant to Stage 1 hypertension | Up to 3 Months
  the blood pressure (mmHg) of people with blood pressures relevant to Stage 1 hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Investigator has left Element Materials Technology
Locations (1):
- Element Materials Technology, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Contactless and Calibration-free Blood Pressure and Pulse Rate Monitor for Screening and Monitoring of Hypertension: Cross-sectional Validation Study — https://preprints.jmir.org/preprint/57241